CLINICAL TRIAL: NCT03804138
Title: Immune Damage and Vaccination in COPD Patients
Acronym: ALTIBPCO
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Other Study IDs: ALTIBPCO; 2018-A01719-46 (Other: ID-RCB)
Record Dates: First submitted 2019-01-11; First posted 2019-01-15 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient: patient with COPD
  Interventions: Other: Anti-influenza and DTp pertussis vaccinations
- control group: patient without COPD
  Interventions: Other: Anti-influenza and DTp pertussis vaccinations

INTERVENTIONS:
Other: Anti-influenza and DTp pertussis vaccinations — Anti-influenza and DTp pertussis vaccinations will be performed during the visit by the clinical research nurse. The vaccine has been prescribed as part of the care either by the patient's physician (pulmonologist or general practitioner).

SUMMARY:
Better understanding of the specificities of the vaccine response in patients with COPD

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) will become the third leading cause of death worldwide in 2020 (3.5 million patients, 16500 deaths in France). Its socio-economic cost is related to the handicap induced by the decline of the respiratory function, as well as to the occurrence of exacerbations, main causes of hospitalization and mortality. Since exacerbations are mostly infectious, a preventive strategy involves routine influenza vaccination. Although it is highly recommended in this population, there is no formal evidence of its effectiveness during COPD. While correlates of influenza vaccine efficacy exist, cellular and humoral responses to this vaccine have been poorly evaluated in these patients. This alteration of the vaccine response could also be integrated into an overall deficit of the response to a vaccine in these patients.

As influenza virus infection is one of the most important causes of death in patients with COPD, and vaccination is the best way to prevent it, it is essential to better understand the immune response in the context of vaccination in this population. The investigator's hypothesis is that there would be a global alteration of the immunological immune response in the COPD patient involving abnormalities of lymphocyte B differentiation and the effector capacity of T lymphocytes, notably through the activation of the PD1 / PDL1 axis.

ELIGIBILITY:
Inclusion Criteria:

* Acceptance to participate in the protocol
* Affiliated to a social security scheme
* Age between 40 and 65 years COPD patients
* Diagnosis of moderate to very severe COPD with FEV1 / FVC <0.7 and FEV1 <80% of predicted value, cumulative smoking greater than 10PA
* Indication reminder dTP pertussis when the last booster <5 years Patients without COPD
* FEV / FVC> 0.8
* Indication reminder dTP pertussis when the last booster <5 years
* Indication and patient's wish for an influenza vaccination

Exclusion Criteria:

* Refusal to participate in the study
* Progressive cancer and / or treated in the last 5 years, uncontrolled heart failure, connective tissue disease, inflammatory disease of the digestive tract during treatment.
* Exacerbation or any upper or lower respiratory infection in the previous month.
* Any cause of immunodepression, including long-term oral corticosteroids.
* Pregnant or lactating woman

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be offered to patients for whom there is a prescription for influenza vaccination and DTp, COPD or non-COPD
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2021-02-03 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
Rate and evolution of specific antibodies and Cellular B vaccine response | 30 days
  Rate and evolution of J30-specific antibodies according to WHO criteria Tetanus: before vaccination a rate> 0.1 IU / ml is considered protective, that is usually at a rate> 1 IU / ml after booster vaccination Influenza: antibody concentrations exceeding 0.15 μg / ml are considered protective Pertussis: anti-pertussis toxin IgG (PT) Cellular B vaccine response (plasmablast on D7)

SECONDARY OUTCOMES:
Type of Cellular T cell response | 15 days
  Cellular T cell response (Tfh, Treg, TCD4 / TCD8 specific)
Transcriptomic analysis | 30 days
  Transcriptomic analysis in the pre- and post-vaccination period (vaccine signature) and comparison with matched subjects
Number of Lymphocyte populations | 7 days
  Analysis of lymphocyte populations B and T
Number of exacerbations | 6 months
  Number of minimal, moderate and severe exacerbations within 6 months of vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Boyer, MD, Principal Investigator — CHU Henri-Mondor
Locations (2):
- France (2):
  - CHI Créteil, Créteil
  - CHU Henri-Mondor, Créteil